## INFORMED CONSENT: PARENT/ LEGAL GUARDIAN

**TITLE:** Acute responses to a potentiation warm-up protocol on sprint and change of direction in female football players: a randomized controlled study

**Date:** 28/03/2023

| Ι, | , identification |
|---|---|
| card/passport number | , parent/legal guardian of the player |
| -, identification card/passport number | |
| participating in the research Project entitled: | "Interindividual variability in response to a |
| potentiation warm-up protocol on sprint and | COD in female soccer players: a randomized |
| controlled study". | |
| This study assumes the creation of two | groups: an experimental group and a control |
| group. The experimental group will be exposed | to a potentiation protocol as a warm-up, while |

This study assumes the creation of two groups: an experimental group and a control group. The experimental group will be exposed to a potentiation protocol as a warm-up, while the control group will perform their usual training warm-up program. The distribution between the experimental and control groups will be done randomly and definitively. All players participating in the study will be subject to the 40-meter sprint test and the agility T-test before and after the application of the study protocol. This intervention will be spread over 3 weeks. The first week will be dedicated to familiarizing the players with the tests and protocol, during which two training sessions will be required for the respective procedures. The following two weeks will be dedicated to collecting test data using the protocol, which will be divided into four training sessions, two training sessions per week.

The only risks. That may be associated with this study are the possible risks inherent in to the practice of football. Even so, the players are protected by the sports insurance that they are entitled to at the Club, and since the exposure to this protocol will take place during a training period, all players are protected in this sense.

Finally, I understand that my daughter's participation is voluntary and that she may choose to withdraw from the study at any time without having to provide any justification. Furthermore, the. Data collected will be anonymized and confidential. However, at a later stage of the study, only the substantial data will be used to explain the results obtained, without mentioning any personal information relating to any participant in this study.

By signing, I confirm that. I have read the above information and that I have had the opportunity to clarify any other associated questions.

| Porto, | de | _de 2023 |
|---|---|---|
| Parent/Legal guardi | ian: | |
| The principal investigator, in the name | of the entire inves | stigation team: |